CLINICAL TRIAL: NCT07157670
Title: Cardiovascular Complications in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation.
Acronym: ALLOCARDIOTOX
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-S 942 MASCOT (Unknown); INSERM U1086 Cancers et Préventions (Unknown); Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250015; N°IDRCB: 2025-A00066-43 (Other: ANSM)
Record Dates: First submitted 2025-08-19; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cardiotoxicity; DPP3; HSCT; Allogeneic Hematopoietic Stem Cell Transplantation; ACS - Acute Coronary Syndrome; Cardiac Dysfunction; Arrythmia, Cardiac; Pulmonary Hypertension; Machine Learning
Keywords: DPP3; HSCT; Cardiotoxicity; Allogeneic hematopoietic stem cell transplantation; Machine Learning
MeSH Terms: conditions — Cardiotoxicity; Acute Coronary Syndrome; Arrhythmias, Cardiac; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Evaluate DPP3 as a predictive biomarker of cardiac dysfunction in a cohort of consecutive HSCT patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of consecutive HSCT patients.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) represents a major therapeutic strategy for malignant hematologic diseases, with the number of procedures steadily increasing in France each year. Conditioning and maintenance regimens carry a risk of both short- and long-term cardiotoxicity, leading to serious cardiovascular events including acute coronary syndrome (ACS), cardiac dysfunction, arrhythmias, pulmonary hypertension, and pericardial effusion. The pathophysiology of cardiotoxicity in HSCT patients remains poorly understood.

It is therefore crucial to investigate underlying mechanisms and identify predictive factors of cardiotoxicity in order to provide appropriate cardiological follow-up and management. Current European Society of Cardiology guidelines recommend routine monitoring of HSCT patients with echocardiography and cardiac biomarkers (NT-proBNP, troponin), although these recommendations are based on small-scale studies. The cardiodepressor factor DPP3 has shown promising results in cardio-oncology, with a causal role in anthracycline-induced cardiac dysfunction. Its role in HSCT-related cardiotoxicity requires further evaluation.

This multicenter study of HSCT recipients will be a valuable resource, enabling a better understanding of the pathophysiology of cardiotoxicity and prognosis. It will highlight imaging (echocardiography, calcium score, supra-aortic Doppler), electrocardiographic, and biological markers (including DPP3) associated with prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years
* Informed about the study and without objection to participation (or with consent from legal guardians)
* Undergoing allogeneic HSCT

Exclusion Criteria:

* Patient not followed up at the participating center
* Pregnant or breastfeeding women
* Patient not affiliated with social security
* Patient under guardianship, curatorship, or legal protection

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients hospitalized for HSCT in the participating centers, meeting eligibility criteria, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Composite cardiotoxicity outcome during follow-up of 1 year, defined as cardiovascular mortality, cardiac dysfunction, acute coronary syndrome, pericarditis, and supraventricular or ventricular arrhythmias. | During follow-up of 1 year